CLINICAL TRIAL: NCT06378021
Title: Post Operative Atrial Fibrillation: Alleviation by Calcium Chloride Injection Into Cardiac Ganglionic Plexus During Coronary Artery Bypass Grafting.
Brief Title: Role of Calcium Chloride Injection in Alleviating Atrial Fibrillation Post CABG
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Nadine Osama Elgarhi, Doctor of pharmacy, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Calcium chloride in CABG
Record Dates: First submitted 2024-03-22; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Calcium chloride; On pump Coronary artery bypass graft
MeSH Terms: conditions — Atrial Fibrillation | interventions — Calcium Chloride; Sodium Chloride; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium chloride injection in ganglionated plexis for Atrial Fibrillation alleviation post CABG (Experimental): The Patients in the intervention arm will be injected with Calcium chloride in the 4 major atrial ganglionated plexis after the by pass is completed.
  Interventions: Drug: Calcium Chloride
- patients who will receive their regular standard of care without calcium chloride injection (Placebo Comparator): A group of patients who will undergo Coronary artery bypass graft surgery will be injected with normal saline in the ganglionic Plexus during Coronary artery bypass graft to act as a comparator to determine if calcium chloride injection alleviate Atrial fibrillation post surgery
  Interventions: Drug: Sodium Chloride 0.9% Inj

INTERVENTIONS:
Drug: Calcium Chloride — 5 % calcium chloride injection in cardiac ganglionic Plexus during On pump Coronary artery bypass graft
  Other Names: 10% ampoules calcium chloride
  Arms: Calcium chloride injection in ganglionated plexis for Atrial Fibrillation alleviation post CABG
Drug: Sodium Chloride 0.9% Inj — 0.9% sodium chloride injection during on pump during Coronary artery bypass graft
  Other Names: Normal saline
  Arms: patients who will receive their regular standard of care without calcium chloride injection

SUMMARY:
This study hypothesize that injecting calcium chloride (CaCl2) into the major atrial ganglionated plexus (GPs) during on pump Coronary artery bypass graft (CABG) can reduce the incidence of Post operative Atrial fibrillation in the first 7 days after surgery.The study is designed to be prospective interventional study two armed RCT for on pump CABG patient.

The intervention arm will be injected with Calcium chloride in the four major atrial ganglionic plexus The control arm will be injected with sodium chloride to determine the effect of Calcium chloride on Post CABG Atrial fibrillation

DETAILED DESCRIPTION:
This study hypothesize that injecting calcium chloride into the major atrial ganglionic plexus (GPs) during On pump Coronary artery bypass graft (CABG) can reduce the incidence of Post operative Atrial fibrillation by calcium-induced autonomic neurotoxicity, the incidence of Post operative Atrial fibrillation can be reduced by suppressing the function of the major atrial GPs and the surrounding neural network that play an important role in initiating Post operative Atrial fibrillation. The study is designed to be prospective interventional study two armed RCT for on pump CABG patient. The plan of work will include dividing the patients into 2 randomized control groups In the intervention group patients will be injected with 5% Calcium chloride in the 4 Major atrial ganglionic plexus The other arm will be Coronary artery bypass graft patients who will be injected with sodium chloride 0.9% to compare the two groups to evaluate to evaluate the effect of Calcium chloride in post CABG atrial fibrillation between the 2 arms of the study.

ELIGIBILITY:
Inclusion Criteria:

1) Patients more than 18 years old 2 ) patients undergoing On pump CABG

Exclusion Criteria:

1. patients >75 years of age
2. Patients with Pre operative Atrial fibrillation
3. Patients with Significant valvular disease

5. Ejection fraction <30% 6. Combined surgery of any kind 7. Congenital heart disease 8. Abnormal severe liver or kidney dysfunction. 9. Patients undergoing Off-pump CABG 10. Poorly controlled hyperthyroidism 11. Refusal to enrollment.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in number of patients who developed Atrial fibrillation | Up to one week from the time of surgery determined by serial ECGs per day
  Compare if calcium chloride injection decrease the percentage of patients who developed Atrial fibrillation in intervention group with those in placebo group

SECONDARY OUTCOMES:
Change in length of hospital stay | Up to the time of patient discharge from the hospital (from the time of post Coronary artery bypass graft surgery)
  investigate if calcium chloride will decrease duration of hospital stay compared with those in the placebo group who are injected with normal saline

CONTACTS AND LOCATIONS:
Overall Officials: Abdelhameed I Ebid, Principal Investigator — Prof
Locations (1):
- Ain shams university, Cairo, Abassia Cairo, Egypt

REFERENCES:
- [Background] Wang H, Zhang Y, Xin F, Jiang H, Tao D, Jin Y, He Y, Wang Q, Po SS. Calcium-Induced Autonomic Denervation in Patients With Post-Operative Atrial Fibrillation. J Am Coll Cardiol. 2021 Jan 5;77(1):57-67. doi: 10.1016/j.jacc.2020.10.049. PMID 33413942